CLINICAL TRIAL: NCT03456635
Title: Improving Perioperative Antimicrobial Prophylaxis by the Use of a Computerized Decision Support System
Acronym: eSATP
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID
Sponsor: University Hospital, Geneva (Other)
Collaborators: Universidade do Porto (Other); University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Américo Agostinho, Clinical Nurse Specialist, University Hospital, Geneva
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-01881
Record Dates: First submitted 2018-02-22; First posted 2018-03-07 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Surgery
Keywords: antimicrobial; prophylaxys; CDSS

STUDY DESIGN:
Intervention Model Description: quasi-experimental study Time-series analysis, with a non-equivalent variable prospective Quality Improvement project
Masking Description: unblinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- usual antimicrobial prophylaxys (No Intervention): standard of care: perioperative antimicrobial prophylaxis without computerized decision support system
- guided antimicrobial prophylaxis (Experimental): perioperative antimicrobial prophylaxis guided by a computerized decision support system
  Interventions: Other: guided antimicrobial prophylaxis

INTERVENTIONS:
Other: guided antimicrobial prophylaxis — During the intervention period, antimicrobial prophylaxis decisions will be guided by a computerized program
  Arms: guided antimicrobial prophylaxis

SUMMARY:
To evaluate the impact of using a computerized decision program on the adequacy of the perioperative antimicrobial prophylaxis

DETAILED DESCRIPTION:
Adequacy rate of surgical antimicrobial prophylaxis, helped by a computerized decision support system, according to the internal guidelines considering the aspects: drug choice, dosing, timing, and re-dosing

ELIGIBILITY:
Inclusion Criteria:

* All elective & emergency surgeries done by neurosurgery, orthopaedics, cardiovascular and digestive specialties made at University Hospitals of Geneva

Exclusion Criteria:

* Patients < 40 kgs

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Adequacy rate of surgical antimicrobial prophylaxis | baseline & 1 year
  Adequacy rate of surgical antimicrobial prophylaxis according to the internal guidelines

SECONDARY OUTCOMES:
Incidence of surgical site infections | baseline & 1 year
  Incidence of surgical site infections in subgroups: hip & knee, colon & rectum, lumbar neurosurgeries and heart surgeries

CONTACTS AND LOCATIONS:
Overall Officials: Americo Agostinho, BSc, Principal Investigator — Clinical nurse specialist
Locations (1):
- University Hospitals of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No